CLINICAL TRIAL: NCT00639574
Title: Interest of Néfopam in the Treatment of Pain During the Intense Ureteral Calculi Uncomplicated in Adults in Emergencies Unit.
Brief Title: Nefopam and Morphine Consumption in the Treatment of Ureteral Calculi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Moustafa Farès, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0030
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Ureteral Calculi, Hyperalgic, Not Complicated
Keywords: Pain, morphine, nefopam, co analgesia, ureteral calculi, emergency
MeSH Terms: conditions — Ureteral Calculi; Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Néfopam — There are two groups :
  * a group N : néfopam
  * a group P : placebo All the patients receive, before randomization, 100 mg of ketoprofen (Profenid) on 20 minutes.

SUMMARY:
The administration of néfopam after initial treatment by kétoproféne, could obtain, in patients remaining pain and classically need morphine, analgesia at least the same as morphine alone. The use of néfopam second line after ketoprofen could reducing (or even eliminating) the need for morphine (and its side effects), allowing a reduction in the length of stay of patients in the emergency unit.

The main objective is to show that the addition of a néfopam initial treatment with the kétoproféne, reduces, in patients with ureteral calculi, the percentage of patients requiring the use of a treatment by morphine.

The secondary objective is to reduce the side effects caused by the morphine, shorten the time to install the appropriate level of analgesia while reducing the risk of failure of the titration morphine, reduce the time spent on titration of morphine and reduce the length of stay patient intake in emergency unit.

DETAILED DESCRIPTION:
The study is prospective, parallel, double-blind, randomized, placebo-controlled analysis with intent to treat. There are 2 groups:

* A group N: néfopam
* A group P: placebo And all the patient receive, before randomization, 100 mg of ketoprofen (Profenid ®) on 20 minutes.

The number of subjects is 52.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 50 years old.
* Admitted to the emergency room for typical ureteral calculi with severe pain (VAS > or = 60), and microscopic hematuria in the strip without signs of urinary complications.
* Preliminary Agreement patient.

Exclusion Criteria:

* Patient disagree.
* Pregnant women (sought by the questioning).
* Fever > 38 ° C.
* Leucocyturie or nitriturie (dipstick).
* Contraindication to ketoprofen.
* Contraindication to néfopam.
* Contraindication to morphine.
* Contraindication linked to drug interactions as mentioned in the Summary of Product Characteristics of the Authorization for placing on the market of Acupan ®.
* Treatment opioid analgesics, nonsteroidal anti-inflammatory or inflammatory or paracetamol in the previous 12 hours.
* Secondary exclusion to a urinary tract infection or systemic.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Need to use morphine as an analgesic scheme (binary yes/no) | As analgesic scheme

SECONDARY OUTCOMES:
Quantity of morphine consumed after titration (mg and number of bolus) | After titration and after administration of placebo or néfopam
Pain (measured by the EVA) after administration of placebo or néfopam | After titration and after administration of placebo or néfopam
Simplified verbal Scale of Satisfaction | After titration and after administration of placebo or néfopam

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Fares, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moustafa F, Liotier J, Mathevon T, Pic D, Perrier C, Schmidt J. Usefulness of nefopam in treating pain of severe uncomplicated renal colics in adults admitted to emergency units: a randomised double-blind controlled trial. The 'INCoNU' study. Emerg Med J. 2013 Feb;30(2):143-8. doi: 10.1136/emermed-2011-200753. Epub 2012 Mar 16. PMID 22427403